CLINICAL TRIAL: NCT02049593
Title: Phase I Trial of BMN 673 and Selected Cytotoxics in Patients With Advanced Solid Tumors
Brief Title: PARP Inhibitor BMN-673 and Temozolomide or Irinotecan Hydrochloride in Treating Patients With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Translational Research in Oncology (Other); BioMarin Pharmaceutical (Industry); Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-001857; NCI-2014-00048 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); TRIO-US GI-07 (Other: Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2014-01-27; First posted 2014-01-30 (Estimated); Last update posted 2022-09-26 (Actual); Status verified 2019-11

CONDITIONS: Metastatic Cancer; Unspecified Adult Solid Tumor
Keywords: protocol specific
MeSH Terms: conditions — Neoplasm Metastasis | interventions — talazoparib; Temozolomide; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (PARP inhibitor BMN-673, temozolomide) (Experimental): Patients receive PARP inhibitor BMN-673 PO QD on days 1-28 and temozolomide PO daily on days1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: PARP inhibitor BMN-673; Drug: temozolomide; Other: pharmacological study; Other: laboratory biomarker analysis
- Arm B (PARP inhibitor BMN-673, irinotecan hydrochloride) (Experimental): Patients receive PARP inhibitor BNM-673 as in Arm A and irinotecan hydrochloride IV on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: PARP inhibitor BMN-673; Drug: irinotecan hydrochloride; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: PARP inhibitor BMN-673 — Given PO
  Other Names: BMN 673; BMN-673
Drug: temozolomide — Given PO
  Other Names: SCH 52365; Temodal; Temodar; TMZ
  Arms: Arm A (PARP inhibitor BMN-673, temozolomide)
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E
  Arms: Arm B (PARP inhibitor BMN-673, irinotecan hydrochloride)
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and the best dose of poly (adenosine diphosphate [ADP]-ribose) polymerase (PARP) inhibitor BMN-673 when given together with temozolomide or irinotecan hydrochloride in treating patients with locally advanced or metastatic solid tumors. PARP inhibitor BMN-673 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and may help temozolomide and irinotecan hydrochloride work better by making tumor cells more sensitive to the drug. Drugs used in chemotherapy, such as temozolomide and irinotecan hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving PARP inhibitor BMN-673 with temozolomide or irinotecan hydrochloride may be an effective treatment for patients with advanced solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability and to estimate the maximum tolerated dose (MTD) of the following combinations in participants with advanced solid tumors: Arm A: BMN 673 (PARP inhibitor BMN-673) and temozolomide; Arm B: BMN 673 and irinotecan (irinotecan hydrochloride).

SECONDARY OBJECTIVES:

I. To evaluate the pharmacokinetics of BMN 673, temozolomide, and irinotecan when BMN 673 is given in combination with temozolomide (Arm A) or irinotecan (Arm B). To assess the effects of temozolomide and irinotecan in Arms A and B respectively on the pharmacokinetics of BMN 673.

II. To evaluate biomarkers that correlate with effect of BMN 673 in combination with temozolomide or irinotecan.

III. To document any anti-tumor activity.

OUTLINE: This is a dose-escalation study of PARP inhibitor BMN-673. Patients are assigned to 1 of 2 treatment arms.

ARM A: Patients receive PARP inhibitor BMN-673 orally (PO) once daily (QD) on days 1-28 and temozolomide PO daily on days1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive PARP inhibitor BNM-673 as in Arm A and irinotecan hydrochloride intravenously (IV) on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented, unresectable, locally advanced or metastatic solid tumor for which no standard therapy is recognized or for which standard therapy has failed
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST, v1.1)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN); if liver function abnormalities are due to hepatic metastasis, then AST and ALT may be =< 5 x ULN
* Total serum bilirubin =< 1.5 x ULN
* Calculated creatinine clearance of >= 40 ml/min; as per Cockcroft-Gault formula
* Hemoglobin >= 9.0 g/dL
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Able to take oral medications
* Willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research-related procedures
* Sexually active patients must be willing to use an acceptable method of contraception such as double barrier contraception during treatment and for 30 days after the last dose of BMN 673
* Females of childbearing potential must have a negative serum pregnancy test at screening

Exclusion Criteria:

* Has not recovered (recovery is defined as National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE version (v)4.03] grade =< 1) from the acute toxicities of previous therapy, except treatment-related alopecia or laboratory abnormalities otherwise meeting the inclusion requirements stated in the inclusion criterion
* Prior treatment with a PARP inhibitor
* Prior allergic reaction or severe intolerance to either irinotecan or temozolomide
* History of central nervous system (CNS) metastasis that are untreated or not stable
* Any antitumor systemic cytotoxic therapies within 28 days prior to enrollment (6 weeks for nitrosoureas or mitomycin-C); prior high-dose chemotherapy with bone marrow or stem cell transplant is excluded
* Is known to have human immunodeficiency virus (HIV) or has active hepatitis C virus (HCV), or active hepatitis B virus (HBV)
* Has had major surgery within 28 days prior to enrollment
* Active gastrointestinal tract disease with malabsorption syndrome
* Requirement for IV alimentation
* Uncontrolled inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
* Symptomatic congestive heart failure (New York Heart Association > class II), unstable angina, or unstable cardiac arrhythmia requiring medication (atrial fibrillation is permitted)
* Use of any investigational product or investigational medical device within 28 days prior to enrollment
* Concurrent disease or condition that would interfere with study participation or safety, such as:

  * Active, clinically significant infection requiring the use of parenteral anti-microbial agents, or grade > 2 by NCI CTCAE (v 4.03) within 14 days prior to enrollment
  * Clinically significant bleeding diathesis or coagulopathy, including known platelet function disorders
  * Non-healing wound, ulcer, or bone fracture
  * Bone marrow disorder including myelodysplasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-06-12 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity graded using the NCI CTCAE v. 4.03 | Up to 28 days

SECONDARY OUTCOMES:
Incidence of adverse events graded by NCI CTCAE v. 4.03 | Up to 12 months
  Characterized by type, frequency, severity, timing, seriousness, and relationship to study therapy.
Levels of PARP inhibitory BMN 673 | Baseline, at 30 and 60 minutes, at 1.5, 2, 3, 4, 6, and 8 hours of day 1 of courses 1 and 2
levels of temozolomide | Baseline, at 30 and 60 minutes, at 1.5, 2, 3, 4, 6, and 8 hours of day 1 of courses 1 and 2
Levels of irinotecan hydrochloride | Baseline, at 30 and 60 minutes, at 1.5, 2, 3, 4, 6, and 8 hours of day 1 of courses 1 and 2
Biomarker levels in blood and tumor tissue | Baseline and Cycle1 Day 21 for participants undergoing biopsy (expansion phase only)
Incidence of laboratory abnormalities graded by NCI CTCAE v. 4.03 | Up to 12 months
  Characterized by type, frequency, severity, timing, seriousness and relationship to study therapy.
Objective tumor response assessed using RECIST v. 1.1 | Up to 12 months
  Sum of partial responses plus complete responses. The proportion of ever achieving a clinical response will be estimated, and an exact one-sided 90% confidence interval will be constructed to identify the likely range for the underlying tumor response rate.
Duration of response | Time of initial response until documented tumor progression, assessed up to 12 months
  The log rank test will be used to examine association between categorical markers and time to disease progression. Cox-proportional hazards regression models will be used to correlate quantitative markers with time to disease progression.
Progression-free survival | Time from enrollment until objective tumor progression or death, assessed up to 12 months
Overall survival (OS) | Time from randomization until death from any cause, up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Zev Wainberg, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, Los Angeles, California, United States